CLINICAL TRIAL: NCT00004809
Title: Phase I Study of Ex Vivo Liver-Directed Gene Therapy for Familial Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pennsylvania (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12011; UPHS-28040
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Familial Hypercholesterolemia
Keywords: familial hypercholesterolemia; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Metabolism, Inborn Errors; Rare Diseases | interventions — Genetic Therapy

INTERVENTIONS:
Procedure: gene therapy

SUMMARY:
OBJECTIVES:

I. Develop an approach for treating patients with homozygous familial hypercholesterolemia using gene therapy with autologous hepatocytes transduced with a normal low-density lipoprotein receptor gene.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Autologous hepatocytes are obtained from a partial hepatectomy and transduced with a recombinant retroviral vector containing the low-density lipoprotein receptor gene. The transduced hepatocytes are infused via the inferior mesenteric vein 3 days following surgery.

Traditional therapy is discontinued for 4 weeks prior to protocol therapy and may resume 6 weeks after the hepatocyte infusion.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Homozygous familial hypercholesterolemia, i.e.: Low-density lipoprotein (LDL) cholesterol greater than 500 mg/dL Autosomal dominant inheritance Early-onset tendon and tuberous xanthomas LDL receptor negative, i.e.: Receptor binding in cultured fibroblasts no more than 20% of normal OR Genotype with 2 previously described, disease-causing alleles Advanced coronary heart disease with relatively poor prognosis, i.e: Angina pectoris History of myocardial infarction Positive exercise tolerance test Atherosclerotic disease in proximal aorta or coronary arteries by ultrasound or angiogram None of the following: Unstable angina pectoris Left ventricular ejection fraction less than 30% Decompensated congestive heart failure Untreated ventricular tachycardia Moderate to severe aortic stenosis Other dyslipidemia Obstructive hepatobiliary disease

* Prior/Concurrent Therapy At least 2 weeks since the following: Drugs affecting cholesterol metabolism Plasma exchange LDL apheresis --Patient Characteristics-- Age: Any age Renal: No azotemia No significant proteinuria Other: No hypothyroidism No diabetes

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1992-06

CONTACTS AND LOCATIONS:
Overall Officials: James M. Wilson, Study Chair — University of Pennsylvania